CLINICAL TRIAL: NCT02042001
Title: A Pilot Randomized Controlled Trial of Switch to Tenofovir Disoproxil Fumarate/Emtricitabine/Rilpivirine (TDF/FTC/RPV) Versus Continue TDF/FTC/Efavirenz (EFV) Treatment Among Virologically Suppressed, HIV-1 Infected Subjects With Mild or Asymptomatic EFV-related Neurocognitive or Neuropsychological Side Effects
Brief Title: Switching From Efavirenz/Atripla to Rilpivirine Among Patients With Neurocognitive or Neuropsychological Side Effects
Acronym: SWEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Giuseppe Lapadula, M.D. Ph.D, Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-IT-264-1331
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-08

CONDITIONS: Impaired Cognition; Depression/Anxiety; Poor Quality Sleep; Quality of Life; HIV-1 Infection
MeSH Terms: conditions — Cognition Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Switch (Experimental): Immediate switch to TDF/FTC/RPV
  Interventions: Drug: Immediate switch to TDF/FTC/RPV
- Deferred Switch (Active Comparator): Switch to TDF/FTC/RPV after 24 weeks
  Interventions: Drug: Switch to TDF/FTC/RPV after 24 weeks

INTERVENTIONS:
Drug: Immediate switch to TDF/FTC/RPV
  Other Names: Eviplera (r)
  Arms: Immediate Switch
Drug: Switch to TDF/FTC/RPV after 24 weeks — Patients will continue current EFV-containing regimen up to week 24 and then will be switched to TDF/FTC/RPV
  Other Names: Eviplera(r)
  Arms: Deferred Switch

SUMMARY:
Despite long-term use in clinical practice, chronic treatment with efavirenz (EFV) has been associated with persistent central nervous system symptoms or mild or even asymptomatic neurocognitive impairment. Whether switching to rilpivirine (RPV) containing regimen is beneficial among patients who experience mild or asymptomatic neurocognitive/neuropsychiatric adverse events during EFV has not been explored yet.

The proposed pilot study will examine whether switching from single tablet regimen TDF/FTC/EFV to single tablet regimen TDF/FTC/RPV is associated with neurocognitive/neuropsychiatric improvement among HIV-infected patients with mild/asymptomatic neurocognitive impairment or neuropsychiatric symptoms during EFV-containing antiretroviral treatment.

Patients under stable treatment with TDF/FTC/EFV, confirmed HIV-1 RNA viral load < 50 copies/mL and altered scores in depression, quality of sleep or anxiety tests and/or alteration in 1 or more domains as assessed by neuropsychological assessment, will be randomized to immediate or deferred (24 weeks) switch to TDF/FTC/RPV. Neurocognitive and neuropsychiatric tests will be repeated after 12, 24 and 48 weeks of follow-up and variations will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ability to sign informed consent
* Continuative treatment with TDF/FTC/EFV for ≥180 days
* HIV-1 RNA viral load < 50 copies/mL in two consecutive determinations (including screening)
* No history of treatment failure and/or evidence of any mutations associated with resistance to NRTI or NNRTI
* No contraindication to treatment with study drugs
* Any one of the following conditions:

  (i) Altered scores in depression, quality of sleep or anxiety tests (ii) Alteration in 1 or more domains as assessed by neuropsychological assessment

Exclusion Criteria:

* Ongoing treatment or predictable need of treatment with proton pump inhibitors
* New AIDS defining condition diagnosed within the 21 days prior to screening
* Previous diagnosis of AIDS dementia complex
* Current alcohol or substance dependence
* Major psychiatric disorders
* Decompensated cirrhosis
* Plasma creatinine >1.2 mg/dl or estimated glomerular filtration rate <60 ml/min (MDRD formula)
* AST, ALT or plasma bilirubin >3 times upper limit of normal
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing/food requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric side effects | 24 weeks
  Proportion of patients with improvement in depression, anxiety or quality of sleep scores, evaluated either as a binary (Yes/No) or on a continuous scale
Neurocognitive side effects | 24 weeks
  - Proportion of patients with improvement in neurocognitive performances in either one of the 7 domains investigated, evaluated either as a binary (Abnormal/Normal) or on a continuous scale (deficit score)
Composite neuropsychiatric/neurocognitive | 24 weeks
  Proportion of patients with improvement in either one of the previous binary end-point (composite end-point)

SECONDARY OUTCOMES:
Symptoms | 24 weeks
  Proportion of patients with self-reported improvement in treatment-related symptoms
Quality of Life | 24 weeks
  Proportion of patients with self-reported improvement in quality of life
Cognitive failure | 24 weeks
  Proportion of patients with improvement in Cognitive Failure Questionnaire
Viral suppression | 12 weeks
  Proportion of patients with HIV-RNA <50 copies/ml after 12 weeks of treatment (ITT-M=F)
Viral failure | 12 weeks
  Proportion of patients with HIV-RNA <400 copies/ml after 12 weeks (ITT-M=F)
Virological efficacy | 24 weeks
  Proportion of patients with HIV-RNA <50 copies/ml after 24 weeks (ITT-M=F)
Safety & Tolerability | 24 weeks
  Proportion of patients discontinuing treatment for intolerance to study drugs or due to side effects

OTHER OUTCOMES:
Resistance | 12 & 24 weeks
  Number of patients with genotypic resistance at failure
Immunological response | 12 & 24 weeks
  Change From Baseline in CD4+ and CD8+ T-Lymphocyte Cell Counts at Weeks 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lapadula, MD, PhD, Principal Investigator — AO San Gerardo of Monza; Andrea Gori, MD, Study Director — AO San Gerardo of Monza
Locations (5):
- Italy (5):
  - Clinic of Infectious Diseases, AO San Gerardo, Monza, MB
  - Spedali Civili - University of Brescia, Brescia
  - Clinica di Malattie Infettive, Ospedale San Martino, Genova
  - AO San Paolo - University of Milan, Milan
  - Ospedale Amedeo di Savoia - University of Turin, Torino